CLINICAL TRIAL: NCT06181864
Title: Emotional Regulation to Manage Anxiety and Anger in Individuals With Autism
Brief Title: Emotional Regulation in Individuals With Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2023-011
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; children; emotional regulation; anxiety
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Emotional Regulation; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Twenty children from the experimental group will undergo the treatment using Robot Nao.
  Interventions: Other: NAO intervention
- Control group (Other): Twenty children belonging to the control group will be subjected to the same training but in a traditional way.
  Interventions: Other: Traditional intervention

INTERVENTIONS:
Other: NAO intervention — The subjects will undergo a pre-intervention assessment phase that will consist of administering the Test of Emotional Vocabulary (TLE) and the Test of emotion comprehension (TEC). The tests will be re-submitted at the end of the intervention. Having ascertained the presence of the inclusion criteria and following randomization of the sample, the Experimental Group constituted of 20 children, will be administered the research task, which involves 15 sessions, one per week lasting one hour and thirty minutes. the children are guided by the voice of the robot Nao. The robot guides them in carrying out practical and relaxation activities. Consequently, audio visual feedback will be provided, via the robot, to return information to the subject about the accuracy of the response.
  Arms: Experimental group
Other: Traditional intervention — The subjects will undergo a pre-intervention assessment phase that will consist of administering the Test of Emotional Vocabulary (TLE) and the Test of emotion comprehension (TEC). The tests will be re-submitted at the end of the intervention. Having ascertained the presence of the inclusion criteria and following randomization of the sample, the Experimental Group constituted of 20 children, will be administered the research task, which involves 15 sessions, one per week lasting one hour and thirty minutes. The children are guided by the instructions of the operator who guides them in carrying out practical and relaxation activities. Consequently, the operator will provide feedback, to return information to the subject regarding the accuracy of the response.
  Arms: Control group

SUMMARY:
The objective of the study is to learn about and manage emotions such as anxiety and anger. The activities are aimed at identifying and managing emotions such as anxiety and anger, through the recognition of the changes that occur at a physiological, cognitive, behavioral and communicative level. In the first sessions, children will be exposed to the emotion of happiness through pleasant activities and involved in relaxation exercises. In subsequent sessions, anger and then anxiety will be addressed first. Social tools will be introduced and ways of thinking and perspective useful to children will be addressed. Furthermore, they will learn to use all the tools and strategies necessary to face and overcome the various emotions and situations in a functional manner. In the final sessions, children will work to design a cognitive-behavioral intervention program for themselves and other group members to improve the management of anxiety and anger. The expected results concern the acquisition of adequate emotional regulation; the construction of functional thoughts, social tools, thinking and perspective tools, adequate strategies for managing emotions; the design of a cognitive-behavioral intervention program in daily life and the strengthening of relational, social, empathic and resilient skills within the peer group and families.

ELIGIBILITY:
Inclusion Criteria:

* Proven diagnosis of autism;
* QS ≥ 75;

Exclusion Criteria:

* presence of other medical disorders

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Anxiety Scale for Children (MASC2) | The estimated time for administration of this sub-test is about 10-15 minutes.
  The Multidimensional Anxiety Scale for Children 2nd Edition (MASC 2™) is a questionnaire for assessing the main dimensions of anxiety in children and adolescents. The scale was constructed using a bottom-up empirical approach to ensure that numerous symptom dimensions were included. The item selection procedure categorized the different dimensions of anxiety into emotional, cognitive, physical and behavioral symptoms. The end result of this process was the creation of a multidimensional measure of childhood anxiety that included four factors (physical symptoms, social anxiety, separation anxiety/panic, and danger avoidance) and six subscales (tension/restlessness, somatic /autonomic, perfectionism, anxious coping, humiliation/rejection and performance anxiety).
Screen for Child Anxiety Related Disorders (SCARED) | The estimated time for administration of this sub-test is about 10-15 minutes.
  The SCARED - Screen for child Anxiety Related Emotional Disorders questionnaire is considered one of the best tools for measuring childhood anxiety. The SCARED is a child and parent self-report instrument used to screen for childhood anxiety disorders including general anxiety disorder, separation anxiety disorder, panic disorder, and social phobia. Also, evaluate symptoms related to school phobias.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Istituto per la Ricerca e l'Innovazione Biomedica
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attwood T. Esplorare i sentimenti, terapia cognitivo comportamentale per gestire ansia e rabbia, Armando Editore 2013
- [Background] Conner CM, White SW, Scahill L, Mazefsky CA. The role of emotion regulation and core autism symptoms in the experience of anxiety in autism. Autism. 2020 May;24(4):931-940. doi: 10.1177/1362361320904217. Epub 2020 Feb 12. PMID 32050774
- [Background] Conner CM, Elias R, Smith IC, White SW. Emotion Regulation and Executive Function: Associations with Depression and Anxiety in Autism. Res Autism Spectr Disord. 2023 Mar;101:102103. doi: 10.1016/j.rasd.2023.102103. Epub 2023 Jan 9. PMID 36741741